CLINICAL TRIAL: NCT00758524
Title: A Multi-center, Randomized, Double-blind, Placebo and Active Controlled, Parallel Group, Dose Finding Study to Evaluate the Efficacy and Safety of LCI699 Compared to Placebo After 8 Weeks Treatment in Patients With Essential Hypertension
Brief Title: A Study to Evaluate Efficacy and Safety of LCI699 in Participants With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCI699A2201
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; Phase 2 study; Antihypertensive agent
MeSH Terms: conditions — Essential Hypertension | interventions — Osilodrostat; Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Core Period: LCI699 0.25 mg QD (Experimental): Participants received LCI699 0.25 mg capsules, orally, once daily (QD), with or without food for up to 8 weeks.
  Interventions: Drug: LCI699
- Core Period: LCI699 0.5 mg QD (Experimental): Participants received LCI699 0.5 mg capsules, orally, QD, with or without food for up to 8 weeks.
  Interventions: Drug: LCI699
- Core Period: LCI699 1.0 mg QD (Experimental): Participants received LCI699 1 mg capsules, orally, QD, with or without food for up to 8 weeks.
  Interventions: Drug: LCI699
- Core Period: LCI699 0.5 mg BID (Experimental): Participants received LCI699 0.5 mg capsules, orally, twice daily (BID), with or without food for up to 8 weeks.
  Interventions: Drug: LCI699
- Core Period: Eplerenone 50 mg BID (Active Comparator): Participants received eplerenone 50 mg capsules, orally, BID, with or without food for up to 8 weeks.
  Interventions: Drug: Eplerenone
- Core Period: Placebo (Placebo Comparator): Participants received LCI699-matching placebo or eplerenone-matching placebo, capsules, orally, QD or BID, with or without food for up to 8 weeks.
  Interventions: Drug: LCI699-matching Placebo; Drug: Eplerenone-matching Placebo
- Withdrawal Period: LCI699 0.25 mg QD (Experimental): Participants received LCI699 0.25 mg capsules, orally, QD, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: LCI699
- Withdrawal Period: LCI699 0.25 mg QD Placebo (Placebo Comparator): Participants received LCI699 matching placebo capsules, orally, QD, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: LCI699-matching Placebo
- Withdrawal Period: LCI699 0.5 mg QD (Experimental): Participants received LCI699 0.5 mg capsules, orally, QD, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: LCI699
- Withdrawal Period: LCI699 0.5 mg QD Placebo (Placebo Comparator): Participants received LCI699 matching placebo capsules, orally, QD, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: LCI699-matching Placebo
- Withdrawal Period: LCI699 1.0 mg QD (Experimental): Participants received LCI699 1 mg capsules, orally, QD, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: LCI699
- Withdrawal Period: LCI699 1.0 mg QD Placebo (Placebo Comparator): Participants received LCI699 matching placebo capsules, orally, QD, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: LCI699-matching Placebo
- Withdrawal Period: LCI699 0.5 mg BID (Experimental): Participants received LCI699 0.5 mg capsules, orally, BID, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: LCI699
- Withdrawal Period: LCI699 0.5 mg BID Placebo (Placebo Comparator): Participants received LCI699 matching placebo capsules, orally, BID, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: LCI699-matching Placebo
- Withdrawal Period: Eplerenone 50 mg BID (Active Comparator): Participants received eplerenone 50 mg capsules, orally, BID, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: Eplerenone
- Withdrawal Period: Eplerenone 50 mg BID Placebo (Placebo Comparator): Participants received eplerenone matching placebo capsules, orally, BID, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: Eplerenone-matching Placebo
- Withdrawal Period: Placebo (Placebo Comparator): Participants received LCI699-matching placebo or eplerenone-matching placebo, capsules, orally, QD or BID, with or without food for up to 1 week (Week 8 to Week 9).
  Interventions: Drug: LCI699-matching Placebo; Drug: Eplerenone-matching Placebo

INTERVENTIONS:
Drug: LCI699 — LCI699 oral capsules
  Arms: Core Period: LCI699 0.25 mg QD; Core Period: LCI699 0.5 mg BID; Core Period: LCI699 0.5 mg QD; Core Period: LCI699 1.0 mg QD; Withdrawal Period: LCI699 0.25 mg QD; Withdrawal Period: LCI699 0.5 mg BID; Withdrawal Period: LCI699 0.5 mg QD; Withdrawal Period: LCI699 1.0 mg QD
Drug: Eplerenone — Eplerenone oral capsules
  Arms: Core Period: Eplerenone 50 mg BID; Withdrawal Period: Eplerenone 50 mg BID
Drug: LCI699-matching Placebo — LCI699-matching placebo oral capsules
  Arms: Core Period: Placebo; Withdrawal Period: LCI699 0.25 mg QD Placebo; Withdrawal Period: LCI699 0.5 mg BID Placebo; Withdrawal Period: LCI699 0.5 mg QD Placebo; Withdrawal Period: LCI699 1.0 mg QD Placebo; Withdrawal Period: Placebo
Drug: Eplerenone-matching Placebo — Eplerenone-matching placebo oral capsules
  Arms: Core Period: Placebo; Withdrawal Period: Eplerenone 50 mg BID Placebo; Withdrawal Period: Placebo

SUMMARY:
This study was a proof-of-efficacy, dose finding study of LCI699 in participants with mild-to-moderate uncomplicated essential hypertension in order to assess the blood pressure (BP) lowering effect, safety and tolerability of LCI699 as compared to placebo and eplerenone.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-fertile females.
* 18-75 years inclusive.
* Participants with mild-to-moderate uncomplicated essential hypertension.

Exclusion Criteria:

* All women of child bearing potential.
* Female participants on hormone replacement therapy.
* Severe hypertension.
* History or evidence of a secondary form of hypertension.
* Known moderate or malignant retinopathy.
* History of angina pectoris, myocardial infarction, coronary bypass surgery,ischemic heart disease, surgical or percutaneous arterial intervention of any kind (coronary, carotid or peripheral vessels), stroke, transient ischemic attack (TIA), carotid artery stenosis, aortic aneurysm or peripheral arterial disease.
* Type 1 or type 2 diabetes mellitus.
* Clinically significant valvular heart disease.
* Congestive heart failure (New York Heart Association [NYHA] class II-IV).
* Cardiac electrical abnormalities indicating significant risk of safety for participant taking part in the study.
* History of malignancy of any organ system, treated or untreated, within the past 5 years.
* Liver disease such as cirrhosis or chronic active hepatitis.
* Any surgical or medical conditions that may significantly alter the absorption, distribution, metabolism or excretion of any drug substance
* Any surgical or medical conditions, not identified in the protocol that in the opinion of the investigator or the monitor, place the participant at higher risk from his/her participation in the study, or is likely to prevent the participant from complying with the requirements of the study or completing the trial period.
* Participant unwilling or not able to discontinue safely the use of current antihypertensive medications during the study period
* Any contraindication or history of hypersensitivity to any of the study drugs or to drugs with similar chemical structures.
* Chronic oral or parenteral corticosteroid treatment.
* Treatment with potassium supplement or potassium sparing diuretics.
* Treatment with potent cytochrome P450 3A4 (CYP3A4) inhibitors during the study period.
* Use of other investigational drugs at Visit 1, or within 30 days or 5 half-lives of Visit 1, whichever is longer, unless local health authority guidelines mandate a longer period.
* Serum potassium > 5.2 milliequivalents per liter (mEq/L) or < 3.5 mEq/L at Visit 1.
* Serum sodium < 132 mEq/L at Visit 1.
* Aspartate aminotransferase (ALT) or alanine aminotransferase (AST) > 2 times the upper limit of the normal range (ULN) at Visit 1.
* Bilirubin (total) > 1.5 x ULN at Visit 1.
* Modification of diet in renal disease estimated glomerular filtration rate (MDRD eGFR) < 60 milliliters per minute (ml/min)/1.73 m^2 at Visit 1.
* Other clinically significant laboratory abnormalities, confirmed by repeat measurements, at Visit 1.
* History of active substance abuse (including alcohol).
* Participants with night-shift employment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2008-09-11 (Actual); Primary Completion 2009-07-02 (Actual); Study Completion 2009-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Schumacher CD, Steele RE, Brunner HR. Aldosterone synthase inhibition for the treatment of hypertension and the derived mechanistic requirements for a new therapeutic strategy. J Hypertens. 2013 Oct;31(10):2085-93. doi: 10.1097/HJH.0b013e328363570c. PMID 24107737
- [Derived] Calhoun DA, White WB, Krum H, Guo W, Bermann G, Trapani A, Lefkowitz MP, Menard J. Effects of a novel aldosterone synthase inhibitor for treatment of primary hypertension: results of a randomized, double-blind, placebo- and active-controlled phase 2 trial. Circulation. 2011 Nov 1;124(18):1945-55. doi: 10.1161/CIRCULATIONAHA.111.029892. Epub 2011 Oct 10. PMID 21986283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 84 investigative sites in Argentina, Australia, France, Germany, Netherlands, Romania, Spain, Sweden, and the United States from 11 September 2008 to 02 July 2009.
Pre-assignment Details: A total of 628 participants were enrolled in the study. Out of 628, only 524 participants with essential hypertension were randomized to receive LCI699 or eplerenone in comparison with placebo for 8 weeks, followed by a randomized withdrawal period to either continue the treatment arm they were randomized to or to take placebo for one additional week (Week 9).
Period: Core Period (Week 0 to Week 8)
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo | Withdrawal Period: LCI699 0.25 mg QD | Withdrawal Period: LCI699 0.25 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg QD | Withdrawal Period: LCI699 0.5 mg QD Placebo | Withdrawal Period: LCI699 1.0 mg QD | Withdrawal Period: LCI699 1.0 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg BID | Withdrawal Period: LCI699 0.5 mg BID Placebo | Withdrawal Period: Eplerenone 50 mg BID | Withdrawal Period: Eplerenone 50 mg BID Placebo | Withdrawal Period: Placebo
Started | 92 | 88 | 86 | 97 (One participant in this arm group was randomized twice and was excluded from Full Analysis Set.) | 84 | 77 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated (Safety Set included participants who received at least 1 dose of study drug.) | 92 | 87 | 87 (One participant from LCI699 0.5 mg QD was randomized to LCI699 1.0 mg QD and received LCI699 1.0 mg QD, thus was included in this arm in the Safety Set.) | 97 | 84 | 76 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 84 | 81 | 77 | 90 | 75 | 67 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 7 | 9 | 7 | 9 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 2 | 4 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative Problems | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Abnormal Laboratory Values | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Abnormal Test Procedure Results | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Withdrawal Period (Week 8 to Week 9)
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo | Withdrawal Period: LCI699 0.25 mg QD | Withdrawal Period: LCI699 0.25 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg QD | Withdrawal Period: LCI699 0.5 mg QD Placebo | Withdrawal Period: LCI699 1.0 mg QD | Withdrawal Period: LCI699 1.0 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg BID | Withdrawal Period: LCI699 0.5 mg BID Placebo | Withdrawal Period: Eplerenone 50 mg BID | Withdrawal Period: Eplerenone 50 mg BID Placebo | Withdrawal Period: Placebo
Started (Participants that started the withdrawal period included those who received at least one dose of the study drug from Week 8 to Week 9 (Randomized Withdrawal Safety Set).) | 0 | 0 | 0 | 0 | 0 | 0 | 46 | 38 | 44 | 37 (One participant randomized to Placebo arm in Withdrawal Period received LCI699 0.5 mg QD and was counted in LCI699 0.5 mg QD arm in the Randomized Withdrawal Safety Set.) | 41 | 37 (One participant randomized to LCI699 0.5 mg BID in the core period received LCI699 1.0 mg QD and was considered in the LCI699 1.0 mg QD arm in Randomized Withdrawal Safety Set.) | 45 | 45 | 39 | 36 | 66
Randomized Withdrawal Set (Randomized Withdrawal Set included all participants with post-baseline blood pressure measurements from Week 8 to Week 9 only.) | 0 | 0 | 0 | 0 | 0 | 0 | 45 | 38 | 43 | 37 | 41 | 36 | 45 | 44 | 39 | 36 | 67 (One participant randomized to Placebo arm in Withdrawal Period received LCI699 0.5 mg QD and was counted in LCI699 0.5 mg QD arm in the Randomized Withdrawal Safety Set. However, this participant was counted in the Placebo arm (N=67) in the Randomized Withdrawal Set.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 45 | 38 | 42 | 37 | 41 | 37 | 45 | 45 | 39 | 36 | 66
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Therapeutic Effect | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population included all randomized participants or participants that met the inclusion criteria as described in study documentation protocol excluding misrandomized participants or participants with protocol violations.
Groups:
- Core Period: LCI699 0.25 mg QD: Participants received LCI699 0.25 mg capsules, orally, QD, with or without food for up to 8 weeks.
- Core Period: LCI699 0.5 mg BID: Participants received LCI699 0.5 mg capsules, orally, BID, with or without food for up to 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo | Total
Number analyzed (Participants) | 92 | 87 | 86 | 96 | 84 | 77 | 522
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.5) | 54.8 (7.8) | 54.5 (9.7) | 54.4 (10.8) | 55.3 (9.1) | 53.9 (8.7) | 54.5 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 31 | 33 | 28 | 31 | 181
  Male | 63 | 58 | 55 | 63 | 56 | 46 | 341
Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] — Ambulatory blood pressure monitoring (ABPM) measured a participant's blood pressure (BP) over 24-hour period readings using an automated validated monitoring device at Baseline. The 24-hour ambulatory DBP and 24-hour ambulatory SBP were calculated by taking the mean of all ambulatory DBP and SBP readings respectively for the 24-hour period. Population: Only participants with available ABPM measurements were included for assessment of 24-hour ambulatory DBP and 24-hour SBP.
  millimeters of mercury (mm Hg)
    Clinic Systolic Blood Pressure (SBP) | 157.72 (12.163) | 157.04 (11.580) | 159.24 (10.415) | 158.50 (11.028) | 158.20 (10.954) | 156.69 (10.121) | 157.93 (11.074)
    Clinic Diastolic Blood pressure (DBP) | 100.43 (3.884) | 99.94 (3.314) | 100.03 (3.580) | 100.21 (3.450) | 100.39 (3.607) | 100.54 (3.814) | 100.25 (3.599)
    24-hour Ambulatory SBP: number analyzed (Participants) | 79 | 76 | 80 | 78 | 71 | 66 | 450
    24-hour Ambulatory SBP | 141.97 (11.167) | 140.08 (13.502) | 143.85 (11.613) | 142.20 (11.079) | 143.30 (13.989) | 142.07 (13.150) | 142.25 (12.405)
    24-hour Ambulatory DBP: number analyzed (Participants) | 79 | 76 | 80 | 78 | 71 | 66 | 450
    24-hour Ambulatory DBP | 90.13 (8.893) | 89.33 (8.208) | 91.38 (7.998) | 90.81 (8.260) | 91.14 (8.861) | 90.11 (10.439) | 90.49 (8.744)

OUTCOME MEASURES:

1. Primary Outcome: Core Period: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP) at Week 8 Last Observation Carried Forward (LOCF), as Measured by Office Blood Pressure (OBP)
Description: Automated arterial BP determinations were made after the participant was in the sitting position for 5 minutes according to the Guidelines for management of hypertension: report of the 4th working party of the British Hypertension Society, 2004-BHS IV, using an automated BP device (such as the Omron BP monitor). The change in the MSDBP was calculated comparing the Week 8 readings to the readings taken at Baseline. The change from baseline in MSDBP was analyzed using an analysis of covariance model (ANCOVA) with treatment and region as factors and baseline MSDBP level as a covariate.
Time Frame: Baseline, Week 8
Population: FAS population included all randomized participants or participants that met the inclusion criteria as described in study documentation protocol excluding misrandomized participants or participants with protocol violations. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 92 | 85 | 86 | 96 | 84 | 76
mm Hg | -4.47 (0.60) | -5.50 (0.57) | -7.11 (0.88) | -4.25 (0.95) | -7.49 (0.97) | -3.22 (0.87)

2. Secondary Outcome: Core Period: Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP) at Week 8 LOCF, as Measured by OBP
Description: Automated arterial BP determinations were made after the participant was in the sitting position for 5 minutes according to the Guidelines for management of hypertension: report of the 4th working party of the British Hypertension Society, 2004-BHS IV, using an automated BP device (such as the Omron BP monitor). The change in the MSSBP was calculated comparing the Week 8 readings to the readings taken at Baseline. The change from baseline in MSSBP was analyzed using an ANCOVA with treatment and region as factors and baseline MSSBP levels as a covariate.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 92 | 85 | 86 | 96 | 84 | 76
mm Hg | -9.00 (1.40) | -10.69 (0.98) | -11.93 (1.44) | -9.10 (1.45) | -13.31 (1.48) | -2.93 (1.68)

3. Secondary Outcome: Core Period: Number of Participants With Adverse Event (AEs), Serious Adverse Events (SAEs), and Deaths
Description: An AE was an adverse medical event which occurs in a participant of the study and which is not necessarily in a causal relationship with the treatment the participant receives. SAEs were AEs leading to death, are life-threatening, require hospitalizations or prolongation of hospitalizations, represent an innate malformation or a congenital abnormality.
Time Frame: AEs: From start of the study drug treatment up to 8 weeks; SAE: From signing of the informed consent up to 8 weeks
Population: Safety Set included all the participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 92 | 87 | 87 | 97 | 84 | 76
Participants
  AEs | 23 | 22 | 24 | 27 | 26 | 23
  SAEs | 1 | 0 | 0 | 0 | 0 | 1
  Deaths | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Core Period: Dose Response Relationship of LCI699 as Measured by Change From Baseline in MSDBP at Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID
Number analyzed (Participants) | 92 | 85 | 86 | 96
mm Hg | -4.47 (0.60) | -5.50 (0.57) | -7.11 (0.88) | -4.25 (0.95)

5. Secondary Outcome: Core Period: Dose Response Relationship of LCI699 as Measured by Change From Baseline in MSSBP at Week 8
Description: as for outcome 2
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID
Number analyzed (Participants) | 92 | 85 | 86 | 96
mm Hg | -9.00 (1.40) | -10.69 (0.98) | -11.93 (1.44) | -9.10 (1.45)

6. Secondary Outcome: Core Period: Change From Baseline in Mean 24 Hour Ambulatory SBP at Week 8 as Measured by Ambulatory Blood Pressure Monitoring (ABPM)
Description: An ABPM measured a participant's BP over a 24-hour period readings using an automated validated monitoring device from Baseline to Week 8. The 24-hour SBP was calculated by taking the mean of all ambulatory SBP readings for the 24-hour period.
Time Frame: Baseline, Week 8
Population: FAS population included all randomized participants or participants that met the inclusion criteria as described in study documentation protocol excluding misrandomized participants or participants with protocol violations. Overall number of participants signifies the number of participants in the FAS who have a Baseline and a Week 8 mean 24-hour ABPM sitting SBP assessment.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 62 | 59 | 68 | 70 | 57 | 52
mm Hg | -7.15 (1.20) | -4.90 (1.22) | -7.73 (1.13) | -6.18 (1.14) | -10.52 (1.25) | 1.11 (1.30)

7. Secondary Outcome: Core Period: Change From Baseline in Mean 24 Hour Ambulatory DBP at Week 8, as Measured by ABPM
Description: An ABPM measured a participant's BP over a 24-hour period readings using an automated validated monitoring device from Baseline to Week 8. The 24-hour DBP was calculated by taking the mean of all ambulatory DBP readings for the 24-hour period.
Time Frame: Baseline, Week 8
Population: FAS population included all randomized participants or participants that met the inclusion criteria as described in study documentation protocol excluding misrandomized participants or participants with protocol violations. Overall number of participants signifies the number of participants in the FAS who have a Baseline and a Week 8 mean 24-hour ABPM sitting DBP assessment.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 62 | 59 | 68 | 70 | 57 | 52
mm Hg | -4.03 (0.91) | -2.44 (0.92) | -4.96 (0.86) | -2.75 (0.86) | -6.03 (0.94) | 1.03 (0.99)

8. Secondary Outcome: Core Period: Trough to Hour Ratio for Change From Baseline in 24-hour Mean Ambulatory DBP at Week 8
Description: Trough to peak ratios were derived from an ANCOVA model containing treatment, region, hour, treatment by hour interaction as factors with Baseline as a covariate.
Time Frame: Baseline, every hour up to 24 hours post-dose at Week 8
Population: FAS population included all randomized participants or participants that met the inclusion criteria as described in study documentation protocol excluding misrandomized participants or participants with protocol violations.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 92 | 87 | 86 | 96 | 84 | 77
ratio
  Week 8, Hour 1 | 3.91 (1.466) | 2.95 (1.541) | 0.27 (1.389) | 3.87 (1.404) | 0.17 (1.544) | 7.11 (1.588)
  Week 8, Hour 2 | 1.44 (1.452) | 1.85 (1.488) | 0.17 (1.397) | 3.44 (1.381) | -1.65 (1.529) | 6.28 (1.586)
  Week 8, Hour 3 | 1.16 (1.477) | 1.13 (1.502) | -0.36 (1.387) | 4.01 (1.369) | -2.42 (1.528) | 4.99 (1.585)
  Week 8, Hour 4 | 0.51 (1.452) | 2.91 (1.488) | 0.35 (1.386) | 2.64 (1.378) | -1.39 (1.541) | 7.02 (1.584)
  Week 8, Hour 5 | 1.11 (1.463) | -0.02 (1.513) | -1.69 (1.385) | 1.45 (1.377) | -2.91 (1.514) | 4.31 (1.584)
  Week 8, Hour 6 | -1.18 (1.451) | -2.36 (1.487) | -3.01 (1.386) | 1.20 (1.367) | -4.86 (1.513) | 1.82 (1.585)
  Week 8, Hour 7 | -1.85 (1.463) | -0.95 (1.487) | -2.63 (1.406) | 1.21 (1.366) | -3.70 (1.513) | 3.62 (1.599)
  Week 8, Hour 8 | -3.01 (1.464) | -1.38 (1.487) | -2.43 (1.396) | 2.09 (1.366) | -2.30 (1.514) | 2.65 (1.616)
  Week 8, Hour 9 | -1.24 (1.464) | -0.07 (1.487) | -2.25 (1.386) | 3.27 (1.366) | -2.81 (1.515) | 3.30 (1.600)
  Week 8, Hour 10 | -0.59 (1.452) | 2.60 (1.487) | -1.65 (1.385) | 0.49 (1.378) | -2.43 (1.515) | 3.86 (1.585)
  Week 8, Hour 11 | -1.02 (1.451) | 1.72 (1.487) | -1.54 (1.386) | 1.54 (1.367) | -1.93 (1.514) | 2.38 (1.585)
  Week 8, Hour 12 | -1.60 (1.451) | 2.53 (1.487) | -3.10 (1.385) | -1.06 (1.367) | -3.20 (1.527) | 3.24 (1.584)
  Week 8, Hour 13 | -4.32 (1.451) | -1.20 (1.487) | -5.31 (1.385) | -1.45 (1.366) | -5.35 (1.513) | 1.52 (1.584)
  Week 8, Hour 14 | -6.47 (1.451) | -3.29 (1.487) | -7.38 (1.385) | -2.96 (1.376) | -7.64 (1.513) | -0.90 (1.584)
  Week 8, Hour 15 | -8.34 (1.452) | -5.82 (1.488) | -8.89 (1.386) | -6.10 (1.377) | -9.03 (1.527) | -1.01 (1.586)
  Week 8, Hour 16 | -8.92 (1.465) | -8.37 (1.491) | -10.50 (1.387) | -9.54 (1.369) | -12.55 (1.528) | -1.61 (1.587)
  Week 8, Hour 17 | -10.26 (1.454) | -10.99 (1.492) | -12.71 (1.398) | -10.38 (1.380) | -12.88 (1.516) | -4.20 (1.604)
  Week 8, Hour 18 | -10.68 (1.456) | -11.73 (1.492) | -11.88 (1.389) | -11.85 (1.379) | -13.49 (1.529) | -6.89 (1.587)
  Week 8, Hour 19 | -10.13 (1.456) | -10.12 (1.493) | -9.74 (1.388) | -10.78 (1.369) | -10.13 (1.517) | -5.84 (1.587)
  Week 8, Hour 20 | -10.73 (1.454) | -8.06 (1.504) | -10.43 (1.408) | -10.49 (1.369) | -10.47 (1.516) | -5.21 (1.602)
  Week 8, Hour 21 | -9.31 (1.453) | -7.68 (1.489) | -9.66 (1.386) | -8.22 (1.377) | -10.51 (1.514) | -4.12 (1.586)
  Week 8, Hour 22 | -7.90 (1.452) | -4.93 (1.487) | -5.37 (1.385) | -6.35 (1.386) | -7.60 (1.513) | -1.09 (1.585)
  Week 8, Hour 23 | -4.94 (1.475) | -1.93 (1.487) | -1.18 (1.385) | -2.67 (1.377) | -5.54 (1.513) | 1.82 (1.599)
  Week 8, Hour 24 | -0.21 (1.477) | 1.45 (1.501) | 0.29 (1.397) | 1.36 (1.370) | -2.78 (1.529) | 1.98 (1.617)

9. Secondary Outcome: Core Period: Trough to Hour Ratio for Change From Baseline in 24-hour Mean Ambulatory SBP at Week 8
Description: as for outcome 8
Time Frame: Baseline, every hour up to 24 hours post-dose at Week 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 92 | 87 | 86 | 96 | 84 | 77
ratio
  Week 8, Hour 1 | -0.54 (1.767) | 0.09 (1.859) | -4.51 (1.674) | -1.42 (1.690) | -5.33 (1.863) | 8.23 (1.915)
  Week 8, Hour 2 | -1.59 (1.752) | 0.15 (1.795) | -3.56 (1.685) | -0.57 (1.663) | -5.90 (1.844) | 6.48 (1.913)
  Week 8, Hour 3 | -2.11 (1.781) | -1.53 (1.811) | -4.86 (1.672) | 0.91 (1.649) | -5.89 (1.843) | 4.60 (1.912)
  Week 8, Hour 4 | -2.06 (1.752) | -1.18 (1.794) | -4.15 (1.672) | 1.50 (1.661) | -5.12 (1.859) | 4.68 (1.912)
  Week 8, Hour 5 | -4.29 (1.766) | -3.09 (1.825) | -3.47 (1.671) | -1.70 (1.660) | -7.22 (1.826) | 2.78 (1.912)
  Week 8, Hour 6 | -4.21 (1.751) | -3.12 (1.794) | -5.88 (1.672) | -1.02 (1.648) | -7.91 (1.826) | 1.42 (1.912)
  Week 8, Hour 7 | -4.95 (1.766) | -2.10 (1.794) | -5.40 (1.697) | -0.76 (1.649) | -8.70 (1.826) | 2.25 (1.930)
  Week 8, Hour 8 | -5.28 (1.766) | -4.69 (1.794) | -5.30 (1.684) | -3.02 (1.649) | -8.06 (1.827) | 3.76 (1.950)
  Week 8, Hour 9 | -3.98 (1.766) | -1.59 (1.795) | -4.78 (1.672) | -1.87 (1.649) | -7.46 (1.828) | 2.39 (1.931)
  Week 8, Hour 10 | -3.69 (1.752) | -0.30 (1.794) | -3.40 (1.672) | -1.73 (1.662) | -7.35 (1.828) | 2.54 (1.913)
  Week 8, Hour 11 | -2.47 (1.751) | -0.43 (1.795) | -4.22 (1.672) | -1.74 (1.649) | -5.75 (1.827) | 3.51 (1.913)
  Week 8, Hour 12 | -5.19 (1.752) | 0.73 (1.794) | -4.35 (1.671) | -3.92 (1.650) | -6.25 (1.843) | 4.69 (1.912)
  Week 8, Hour 13 | -6.45 (1.751) | -2.30 (1.794) | -7.25 (1.671) | -4.05 (1.649) | -8.81 (1.826) | 3.20 (1.912)
  Week 8, Hour 14 | -7.37 (1.751) | -5.68 (1.794) | -9.33 (1.671) | -6.12 (1.660) | -10.91 (1.826) | 0.75 (1.912)
  Week 8, Hour 15 | -10.61 (1.752) | -8.28 (1.795) | -11.26 (1.672) | -9.78 (1.661) | -12.04 (1.842) | 0.02 (1.912)
  Week 8, Hour 16 | -11.71 (1.767) | -10.01 (1.797) | -12.63 (1.672) | -13.03 (1.651) | -16.68 (1.843) | -0.33 (1.914)
  Week 8, Hour 17 | -13.71 (1.754) | -11.96 (1.799) | -15.46 (1.685) | -13.72 (1.664) | -19.59 (1.828) | -3.03 (1.933)
  Week 8, Hour 18 | -14.49 (1.756) | -14.37 (1.800) | -14.54 (1.675) | -15.60 (1.664) | -18.55 (1.844) | -6.35 (1.915)
  Week 8, Hour 19 | -13.78 (1.756) | -13.08 (1.801) | -12.85 (1.674) | -15.93 (1.652) | -15.49 (1.830) | -6.98 (1.914)
  Week 8, Hour 20 | -13.92 (1.756) | -13.22 (1.814) | -12.54 (1.699) | -15.47 (1.652) | -16.09 (1.829) | -6.53 (1.934)
  Week 8, Hour 21 | -14.33 (1.754) | -10.06 (1.797) | -12.78 (1.672) | -13.63 (1.662) | -15.34 (1.827) | -3.89 (1.914)
  Week 8, Hour 22 | -13.46 (1.752) | -8.35 (1.794) | -7.52 (1.671) | -10.55 (1.673) | -12.47 (1.826) | -0.94 (1.912)
  Week 8, Hour 23 | -7.88 (1.780) | -6.23 (1.794) | -5.77 (1.671) | -6.73 (1.661) | -9.02 (1.826) | 2.18 (1.930)
  Week 8, Hour 24 | -3.16 (1.781) | -0.64 (1.810) | -3.45 (1.685) | -3.76 (1.651) | -8.90 (1.844) | 0.70 (1.951)

10. Secondary Outcome: Core Period: Change From Baseline in Plasma Aldosterone Levels at Week 8
Description: Change from baseline was analyzed using plasma aldosterone values measured at Baseline and Week 8.
Time Frame: Baseline, Week 8
Population: Safety Set included all the participants who received at least 1 dose of study drug. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 71 | 69 | 70 | 76 | 64 | 54
picomoles per liter (pmol/L) | -21.5 (122) | -20.0 (156) | -9.9 (266) | -47.5 (170) | 277.1 (429) | -28.8 (163)

11. Secondary Outcome: Core Period: Percentage of Participants With a MSDBP Response and MSDBP Control at Week 8 LOCF
Description: MSDBP response was defined as the percentage of participants with a MSDBP <90 mmHg or a >=10 mmHg reduction from Baseline. MSDBP control was defined as the percentage of participants with a MSDBP <90 mmHg.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 92 | 85 | 86 | 96 | 84 | 76
percentage of participants
  MSDBP Response | 39.1 | 34.1 | 50.0 | 34.4 | 48.8 | 27.6
  MSDBP Control | 32.6 | 29.4 | 41.9 | 29.2 | 45.2 | 18.4

12. Secondary Outcome: Core Period: Percentage of Participants With a MSSBP Response and MSSBP Control at Week 8 LOCF
Description: MSSBP response was defined as the percentage of participants with a MSSBP <140 mmHg or a >=20 mmHg reduction from baseline reduction from baseline. MSSBP control was defined as the percentage of participants with a MSSBP <140 mmHg.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 92 | 85 | 86 | 96 | 84 | 76
percentage of participants
  MSSBP Response | 39.1 | 37.6 | 48.8 | 34.4 | 52.4 | 17.1
  MSSBP Control | 31.5 | 27.1 | 40.7 | 25.0 | 44.0 | 15.8

13. Secondary Outcome: Core Period: Change From Baseline in Plasma Cortisol Levels by Adrenocorticotropic Hormone (ACTH) Stimulation Test
Description: The ACTH stimulation cortisol test was a standard procedure to measure the ability of adrenal cortex to respond to exogenous ACTH and directly assess the adrenal reserve. Serum cortisol concentrations at 1 hour after injection were measured to assess the maximum stimulated cortisol level achieved. Potential adrenal suppression was indicated if the serum cortisol concentration was <500 nanomoles per liter (nmol/L) at 1 hour after the injection.
Time Frame: Baseline, 1 hour post-dose at Week 8
Population: ACTH subset population included all participants prior to treatment with LCI699 and at the end of the treatment interval (Week 8). Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure at the given timepoint
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo
Number analyzed (Participants) | 20 | 23 | 28 | 24 | 22 | 17
nanomoles per liter (nmol/L) | 729.20 (123.753) | 692.74 (117.645) | 604.46 (125.017) | 609.21 (107.923) | 802.32 (134.497) | 822.65 (116.041)

14. Secondary Outcome: Withdrawal Period: Change From Week 8 to Week 9 in MSDBP at Week 9, as Measured by OBP
Description: Automated arterial BP determinations were made after the participant was in the sitting position for 5 minutes according to the Guidelines for management of hypertension: report of the 4th working party of the British Hypertension Society, 2004-BHS IV, using an automated BP device (such as the Omron BP monitor). The change in the MSDBP was calculated comparing the Week 9 readings to the readings taken at Week 8 (Baseline). The change from Week 8 to week 9 in MSDBP was analyzed using an ANCOVA with treatment and region as factors and Week 8 MSDBP level as a covariate.
Time Frame: From Week 8 to Week 9
Population: Randomized Withdrawal Set included all participants with post-baseline blood pressure measurements from Week 8 to Week 9 only. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Withdrawal Period: LCI699 0.25 mg QD | Withdrawal Period: LCI699 0.25 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg QD | Withdrawal Period: LCI699 0.5 mg QD Placebo | Withdrawal Period: LCI699 1.0 mg QD | Withdrawal Period: LCI699 1.0 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg BID | Withdrawal Period: LCI699 0.5 mg BID Placebo | Withdrawal Period: Eplerenone 50 mg BID | Withdrawal Period: Eplerenone 50 mg BID Placebo | Withdrawal Period: Placebo
Number analyzed (Participants) | 45 | 38 | 43 | 37 | 41 | 36 | 45 | 44 | 39 | 36 | 67
mm Hg | 0.5 (0.99) | 0.5 (1.08) | 1.6 (1.01) | -0.2 (1.09) | -0.5 (1.03) | 2.5 (1.11) | 1.3 (1.00) | 1.3 (1.02) | -1.2 (1.06) | 0.4 (1.11) | 1.6 (0.83)

15. Secondary Outcome: Withdrawal Period: Change From Week 8 to Week 9 in MSSBP at Week 9 as Measured by OBP
Description: Automated arterial BP determinations were made after the participant was in the sitting position for 5 minutes according to the Guidelines for management of hypertension: report of the 4th working party of the British Hypertension Society, 2004-BHS IV, using an automated BP device (such as the Omron BP monitor). The change in the MSSBP was calculated comparing the Week 9 readings to the readings taken at Week 8 (Baseline). The change from Week 8 to week 9 in MSSBP was analyzed using an ANCOVA with treatment and region as factors and Week 8 MSSBP level as a covariate.
Time Frame: From Week 8 to Week 9
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Withdrawal Period: LCI699 0.25 mg QD | Withdrawal Period: LCI699 0.25 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg QD | Withdrawal Period: LCI699 0.5 mg QD Placebo | Withdrawal Period: LCI699 1.0 mg QD | Withdrawal Period: LCI699 1.0 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg BID | Withdrawal Period: LCI699 0.5 mg BID Placebo | Withdrawal Period: Eplerenone 50 mg BID | Withdrawal Period: Eplerenone 50 mg BID Placebo | Withdrawal Period: Placebo
Number analyzed (Participants) | 45 | 38 | 43 | 37 | 41 | 36 | 45 | 44 | 39 | 36 | 67
mm Hg | 0.3 (1.66) | 3.3 (1.80) | 0.5 (1.69) | 2.5 (1.82) | 0.4 (1.72) | 5.3 (1.85) | 1.6 (1.68) | 4.4 (1.69) | -1.5 (1.79) | 2.7 (1.86) | 1.8 (1.39)

ADVERSE EVENTS:
Time Frame: AEs: From start of the study drug treatment up to 9 weeks; SAE: From signing of the informed consent up to 9 weeks
Description: Core Period: Safety Set included all the participants who received at least 1 dose of study drug. One participant from LCI699 0.5 mg QD was randomized to LCI699 1.0 mg QD and received LCI699 1.0 mg QD, thus was included in this arm in the Safety Set. Withdrawal period: Randomized Withdrawal Safety Set included participants who received at least one dose of the study drug from Week 8 to Week 9.
Groups:
- Withdrawal Period: Eplerenone 50 mg BID Placebo: Participants received eplerenone-matching placebo capsules, orally, BID, with or without food for up to 1 week (Week 8 to Week 9).
Arm/Group | Core Period: LCI699 0.25 mg QD | Core Period: LCI699 0.5 mg QD | Core Period: LCI699 1.0 mg QD | Core Period: LCI699 0.5 mg BID | Core Period: Eplerenone 50 mg BID | Core Period: Placebo | Withdrawal Period: LCI699 0.25 mg QD | Withdrawal Period: LCI699 0.25 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg QD | Withdrawal Period: LCI699 0.5 mg QD Placebo | Withdrawal Period: LCI699 1.0 mg QD | Withdrawal Period: LCI699 1.0 mg QD Placebo | Withdrawal Period: LCI699 0.5 mg BID | Withdrawal Period: LCI699 0.5 mg BID Placebo | Withdrawal Period: Eplerenone 50 mg BID | Withdrawal Period: Eplerenone 50 mg BID Placebo | Withdrawal Period: Placebo
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/87 | 0/87 | 0/97 | 0/84 | 0/76 | 0/46 | 0/38 | 0/44 | 0/37 | 0/41 | 0/37 | 0/45 | 0/45 | 0/39 | 0/36 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/92 | 0/87 | 0/87 | 0/97 | 0/84 | 1/76 | 0/46 | 0/38 | 0/44 | 0/37 | 0/41 | 0/37 | 0/45 | 0/45 | 0/39 | 0/36 | 0/66
Other Adverse Events (participants affected / at risk) | 22/92 | 22/87 | 24/87 | 27/97 | 26/84 | 23/76 | 2/46 | 1/38 | 1/44 | 0/37 | 3/41 | 5/37 | 4/45 | 3/45 | 2/39 | 0/36 | 3/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Period: LCI699 0.25 mg QD (N=92) | Core Period: LCI699 0.5 mg QD (N=87) | Core Period: LCI699 1.0 mg QD (N=87) | Core Period: LCI699 0.5 mg BID (N=97) | Core Period: Eplerenone 50 mg BID (N=84) | Core Period: Placebo (N=76) | Withdrawal Period: LCI699 0.25 mg QD (N=46) | Withdrawal Period: LCI699 0.25 mg QD Placebo (N=38) | Withdrawal Period: LCI699 0.5 mg QD (N=44) | Withdrawal Period: LCI699 0.5 mg QD Placebo (N=37) | Withdrawal Period: LCI699 1.0 mg QD (N=41) | Withdrawal Period: LCI699 1.0 mg QD Placebo (N=37) | Withdrawal Period: LCI699 0.5 mg BID (N=45) | Withdrawal Period: LCI699 0.5 mg BID Placebo (N=45) | Withdrawal Period: Eplerenone 50 mg BID (N=39) | Withdrawal Period: Eplerenone 50 mg BID Placebo (N=36) | Withdrawal Period: Placebo (N=66)
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Period: LCI699 0.25 mg QD (N=92) | Core Period: LCI699 0.5 mg QD (N=87) | Core Period: LCI699 1.0 mg QD (N=87) | Core Period: LCI699 0.5 mg BID (N=97) | Core Period: Eplerenone 50 mg BID (N=84) | Core Period: Placebo (N=76) | Withdrawal Period: LCI699 0.25 mg QD (N=46) | Withdrawal Period: LCI699 0.25 mg QD Placebo (N=38) | Withdrawal Period: LCI699 0.5 mg QD (N=44) | Withdrawal Period: LCI699 0.5 mg QD Placebo (N=37) | Withdrawal Period: LCI699 1.0 mg QD (N=41) | Withdrawal Period: LCI699 1.0 mg QD Placebo (N=37) | Withdrawal Period: LCI699 0.5 mg BID (N=45) | Withdrawal Period: LCI699 0.5 mg BID Placebo (N=45) | Withdrawal Period: Eplerenone 50 mg BID (N=39) | Withdrawal Period: Eplerenone 50 mg BID Placebo (N=36) | Withdrawal Period: Placebo (N=66)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 3 | 1 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 1 | 2 | 3 | 10 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.